CLINICAL TRIAL: NCT01258023
Title: A Phase II Study to Evaluate the Immunogenicity, Safety and Tolerability of a Seasonal Influenza Vaccine Including H1N1 in Immunocompromised Adults Who Have Undergone Solid Organ Transplantation or Bone Marrow Transplantation and in Age-Matched Healthy Volunteers
Brief Title: Seasonal Flu Vaccine in Adult Transplant Recipients
Acronym: Fluad Tx
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HepNet Study House, German Liverfoundation (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010-022871-78
Record Dates: First submitted 2010-11-18; First posted 2010-12-10 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Immunocompromised; Transplanted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- transplant recipients (Experimental): Immunocompromised Adults Who Have Undergone Solid Organ Transplantation or Bone Marrow Transplantation
  Interventions: Biological: Fluad 1x

INTERVENTIONS:
Biological: Fluad 1x — 15 µg antigen/strain:
  * A/California/07/2009 (H1N1) - like strain
  * A/Perth/16/2009 (H3N2) - like strain
  * B/Brisbane/60/2008- like strain MF59 adjuvant 9.75µg ai 0.5ml

SUMMARY:
The trial investigates the efficacy of adjuvanted seasonal influenza including H1N1 Fluad (R) in immunocompromised adults who have undergone solid organ or bone marrow transplantation. It is expected that when administered once the vaccine fulfills all serological efficacy criteria required for the elderly population age 60 years and older.

ELIGIBILITY:
Inclusion Criteria:

Transplant Recipients:

* Adult subjects 18-60 years of age who have undergone prior renal, cardiac, liver, lung, or bone marrow transplantation for any reason, more than 3 months prior to enrolment
* Patients able to visit the outpatient clinic with a life expectancy of at least one year
* Patients who receive any immunosuppressive treatment currently taken to prevent organ rejection

Healthy Adults:

* Adult subjects 18-60 years of age
* Healthy individuals as determined by medical history, physical assessment and clinical judgment of the investigator
* Within the same age category (+/- 5 years) than the incidental transplanted patient

Transplant Recipients and Healthy Adults:

* Individuals who are able to comply with all study procedures and are available for all clinic visits scheduled in the study
* Women of child-bearing potential (WOCBP) must have used an acceptable contraceptive method for at least 2 months prior to study entry until 3 weeks after vaccination: Female of childbearing potential is defined as a post onset of menarche or pre-menopausal female capable of becoming pregnant. This does not include females who meet any of the following conditions: (1) menopause at least 2 years earlier, (2) tubal ligation at least 1 year earlier, or (3) total hysterectomy
* Acceptable birth control methods are defined as one or more of the following: Hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring, Barrier (condom with spermicide or diaphragm with spermicide) each and every time during intercourse, Intrauterine device (IUD, Monogamous relationship with vasectomized partner. Partner must have been vasectomized for at least six months prior to the subject's study entry

Exclusion Criteria:

* Individuals who received any vaccine within 30 days prior to study entry
* Individuals who received a H1N1 or seasonal influenza vaccination less than 6 months prior to the study
* Influenza diagnosed by a physician within 4 months prior to the study start
* Pregnant or lactating females
* History of an anaphylactic (i.e. life-threatening) reaction to any of the components of the vaccines, including egg and chicken proteins, ovalbumin, kanamycin and neomycin sulphate, formaldehyde and cetyltrimethylammonium bromide (CTAB)
* Subjects who are not able to comprehend and to follow all required study procedures for the whole period of the study
* History of or any current illness that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study
* Temperature is ≥ 38 °C or oral temperature ≥ 38.5 °C within 3 days of intended study vaccination
* Administration of parenteral immunoglobulin compound - including HBIg, blood products, and/or plasma derivatives within 6 months prior to Visit 1 or planned during the full length of the study
* HIV infection, as previously determined or reported
* History of progressive or severe neurological disorders (including Guillain-Barré syndrome and convulsions, but excluding febrile convulsions)
* Subjects participating in another clinical trial and / or receiving investigational drug

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Seroconversion and Seroprotection after 21 days | 21 days
  The observed percentage of seroconversion and seroprotection, as well as the observed GMR (measured by HI) in transplanted patients at day 21 will be compared with the thresholds from the guideline for adults aged over 60 (as outlined above). This study is successful, if all three point estimates pass the corresponding efficacy criteria at day 21. For descriptive purpose two-sided 95%-confidence intervals for the rates and the GMR at day 21 will be presented.

SECONDARY OUTCOMES:
comparison of vaccine efficacy in transplanted versus healthy subjects | 21 and 42 days
  1. The immune response of the H1N1 vaccine is at least as effective in transplanted patients as in the healthy volunteers after one administration. For orientation in the assessment a non-inferiority-margin of 0.45 for the ratio of the geometric mean titers (GMTs) of transplanted patients and age-matched healthy volunteers at day 21 will be used and reflects what can be demonstrated with given sample size.
assessment of primary and secondary outcomes with the two other strains | 21 and 42 days
  The primary and the first main secondary objective will also be evaluated for the other two virus strains (H3N2 and type B) of the trivalent vaccination.
safety issues as number of participants with adverse events | 21 and 42 days and 9 months
  The safety of the study vaccine will be analyzed based on number of subjects exposed to the vaccine with respect to (1) solicited events within 7 days after injection; and (2) non-solicited adverse events at least 21 days after injection. Unsolicited events will include SAEs, AEIs (e.g. neuritis, convulsions, severe allergic reactions, angioedema, non-infectious encephalitis, vasculitis, Guillain-Barrè syndrome, demyelination, Bell's palsy), all other non-solicited AEs, which are routinely collected including onset of chronic diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical School Hannover, Hanover, Germany